CLINICAL TRIAL: NCT03959566
Title: A Phase IIB, Open-Label, Randomized Controlled Dose Ranging Multi-Center Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Exposure-Response Relationship of Different Doses of Sutezolid in Combination With Bedaquiline, Delamanid and Moxifloxacin in Adult Subjects With Newly Diagnosed, Uncomplicated, Smear-Positive, Drug-sensitive Pulmonary Tuberculosis
Brief Title: PanACEA Sutezolid Dose-finding and Combination Evaluation
Acronym: SUDOCU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Sequella, Inc. (Industry); Radboud University Medical Center (Other); University of California, San Francisco (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Prof. Dr., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PanACEA-SUDOCU-01
Record Dates: First submitted 2019-03-11; First posted 2019-05-22 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Tuberculosis; Other Specified Pulmonary Tuberculosis
Keywords: Tuberculosis, Pulmonary; Sutezolid; Randomized Controlled Trial (RCT); PNU-100480; Tuberculosis; Antitubercular Agents; Gram-positive Bacterial Infections; Oxazolidinones; Dose-finding; Combination-evaluation; Safety; Tolerability; Pharmacokinetics (PK); Exposure-Response Relationship; Bedaquiline; Delamanid; Moxifloxacin; Drug-sensitive TB
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis; Gram-Positive Bacterial Infections | interventions — PNU-100480; bedaquiline; OPC-67683; Moxifloxacin; Midazolam

STUDY DESIGN:
Intervention Model Description: 75 participants will be randomized to one of five arms (15 participants per arm) to receive study medication containing bedaquiline, delamanid, and moxifloxacin with different doses of sutezolid, ranging from 0mg sutezolid up to 800mg sutezolid twice a day. Participants will be randomised and stratified by site and HIV status.
  Participants will visit the study clinic on a weekly basis for sputum collection, safety monitoring and receipt of study medication.
  After the completion of three months of experimental treatment participants in the experimental arms will be handed over to government TB programmes to complete their course of anti-TB treatment.
Who Masked: Outcomes Assessor
Masking Description: Laboratory staff, analysing and evaluating the sputum and blood samples of the participants, will be blinded to the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1 (U0) (Active Comparator): Participants receive the following medication for the duration of 12 weeks (with Bedaquiline, Delamanid and Moxifloxacin as per licensed dose):
  * 400 mg Bedaquiline orally once daily for the first 14 days, then 200 mg three times a week.
  * 200 mg Delamanid orally in two daily doses of 100 mg.
  * 400 mg Moxifloxacin orally once daily
  Interventions: Drug: Bedaquiline, Delamanid, Moxifloxacin
- Arm 2 (U600) (Experimental): Participants receive the following medication for the duration of 12 weeks (with Bedaquiline, Delamanid and Moxifloxacin as per licensed dose):
  * 400 mg Bedaquiline orally once daily for the first 14 days, then 200 mg three times a week.
  * 200 mg Delamanid orally in two daily doses of 100 mg.
  * 400 mg Moxifloxacin orally once daily
  * 600 mg Sutezolid orally once daily
  Interventions: Drug: Sutezolid; Drug: Bedaquiline, Delamanid, Moxifloxacin
- Arm 3 (U1200) (Experimental): Participants receive the following medication for the duration of 12 weeks (with Bedaquiline, Delamanid and Moxifloxacin as per licensed dose):
  * 400 mg Bedaquiline orally once daily for the first 14 days, then 200 mg three times a week.
  * 200 mg Delamanid orally in two daily doses of 100 mg.
  * 400 mg Moxifloxacin orally once daily
  * 1200 mg Sutezolid orally once daily
  Interventions: Drug: Sutezolid; Drug: Bedaquiline, Delamanid, Moxifloxacin
- Arm 4 (U600BD) (Experimental): Participants receive the following medication for the duration of 12 weeks (with Bedaquiline, Delamanid and Moxifloxacin as per licensed dose):
  * 400 mg Bedaquiline orally once daily for the first 14 days, then 200 mg three times a week.
  * 200 mg Delamanid orally in two daily doses of 100 mg.
  * 400 mg Moxifloxacin orally once daily
  * 600 mg Sutezolid orally twice daily
  Interventions: Drug: Sutezolid; Drug: Bedaquiline, Delamanid, Moxifloxacin
- Arm 5 (U800BD) (Experimental): Participants receive the following medication for the duration of 12 weeks (with Bedaquiline, Delamanid and Moxifloxacin as per licensed dose):
  * 400 mg Bedaquiline orally once daily for the first 14 days, then 200 mg three times a week.
  * 200 mg Delamanid orally in two daily doses of 100 mg.
  * 400 mg Moxifloxacin orally once daily
  * 800 mg Sutezolid orally twice daily
  * 2 mg Midazolam orally once per day on day-1 and day 14
  Interventions: Drug: Sutezolid; Drug: Bedaquiline, Delamanid, Moxifloxacin; Drug: Midazolam oral solution

INTERVENTIONS:
Drug: Sutezolid — Sutezolid is not licensed yet. Current experience in humans up to Phase IIA. Dose according to randomization to dosing arms 2-5.
  Other Names: PNU-100480
  Arms: Arm 2 (U600); Arm 3 (U1200); Arm 4 (U600BD); Arm 5 (U800BD)
Drug: Bedaquiline, Delamanid, Moxifloxacin — These three licensed drugs form the backbone of a new regimen to which sutezolid is added in arms 2-5.
  Other Names: BDM
Drug: Midazolam oral solution — Midazolam will be administered as per probe drug use in a single dose of 2 mg at day -1 and day 14 to assess the potential of sutezolid for CYP 459 3A4 enzyme induction, as measured by its influence on the ratio of AUCs of the CYP 3A4 probe drug
  Arms: Arm 5 (U800BD)

SUMMARY:
This study is an open-label, randomized, controlled, multi-center Phase IIB dose-finding trial to evaluate the safety, tolerability, pharmacokinetics and exposure-response-relationship of different doses of sutezolid (STZ) in combination with bedaquiline, delamanid and moxifloxacin in adults with newly diagnosed, uncomplicated, smear positive and drug sensitive pulmonary tuberculosis. Participants will be randomized to one of five arms containing bedaquiline, delamanid and moxifloxacin with different doses of STZ (0mg, 600mg once daily (OD), 1200mg OD, 600 mg twice daily (BD), 800 mg BD). Study treatment duration will be three months, followed by a follow-up period of 2 weeks.

The primary objective is to identify the optimal dose of sutezolid to be used in subsequent studies that provides the best efficacy at acceptable safety of the drug by describing the safety, tolerability and exposure toxicity relationship of sutezolid (and its main metabolite) given over three months, in combination with standard-dose bedaquiline, delamanid and moxifloxacin, compared to standard-dose bedaquiline, delamanid and moxifloxacin alone.

DETAILED DESCRIPTION:
This open-label Phase IIB dose-finding, randomized, controlled study with a duration of three months of experimental therapy in adult patients with newly diagnosed, smear positive, uncomplicated, drug sensitive pulmonary tuberculosis (TB) will be carried out to evaluate the safety, efficacy, tolerability, pharmacokinetics and exposure/response-relationship of different doses of sutezolid in combination with bedaquiline, delamanid and moxifloxacin (BDM).

Participants will be randomized to one of five arms containing bedaquiline, delamanid and moxifloxacin with different doses of STZ (0mg, 600mg OD, 1200mg OD, 600 mg BD, 800 mg BD). Study treatment duration will be three month, followed by a follow-up period of 2 weeks.

A total of 75 male or female subjects, aged between 18 and 65 years with newly diagnosed, drug sensitive, uncomplicated, smear-positive, pulmonary TB will be included and randomized to one of five arms containing BDM with different doses of STZ:

* Arm 1 (U0): Bedaquiline, delamanid, moxifloxacin
* Arm 2 (U600): Bedaquiline, delamanid, moxifloxacin, sutezolid 600 mg OD
* Arm 3 (U1200): Bedaquiline, delamanid, moxifloxacin, sutezolid 1200 mg OD
* Arm 4 (U600BD): Bedaquiline, delamanid, moxifloxacin, sutezolid 600 mg BD
* Arm 5 (U800BD): Bedaquiline, delamanid, moxifloxacin, sutezolid 800 mg BD

A sub-study will assess CYP P450 3A4 enzyme induction potential using the probe drug midazolam, given to participants in arm 5.

Using PK data and data from primary efficacy and safety objectives, we will develop an exposure-response and a population PK-model for sutezolid and its main metabolite to support the main objective, selection of a dose for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures including HIV testing.
2. Male or female, aged between 18 and 65 years, inclusive.
3. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
4. Newly diagnosed, previously untreated, drug susceptible pulmonary TB: presence of MDR-TB complex and rapid molecular tests result confirming susceptibility to Rifampicin (RIF) and Isoniazid (INH) such as GeneXpert and/or HAIN MTBDR plus.
5. A chest X-ray (no older than 2 weeks) which, in the opinion of the Investigator, is consistent with TB.
6. Sputum positive on microscopy from concentrated sputum for acid-fast bacilli on at least one sputum sample (at least 1+ on the International Union Against Tuberculosis and Lung Disease (IUATLD) /WHO scale).
7. The participant is willing to forgo consumption of foods high in tyramine for the period of taking study medication
8. The participant is either unable to conceive/father children AND/OR his/her partner is unable to conceive/father children AND/OR they will be using effective methods of contraception, as defined below:

   a. Non-childbearing potential: i. Female participant/sexual partner of male participant - bilateral oophorectomy, and/or hysterectomy or bilateral tubal ligation more than 12 months ago and/or has been postmenopausal with a history of no menses for at least 12 consecutive months ii. Male participant/sexual partner of female participant - vasectomised or has had a bilateral orchidectomy minimally three months prior to screening b. Effective contraception methods: i. Female participants: two methods, including methods that the patient's sexual partner(s) use. At least one must be a barrier method. Contraception must be practised for at least until 12 weeks after the last dose of STZ.

(Note: hormone-based contraception alone may not be reliable when taking RIF during continuation Phase; therefore, hormone-based contraceptives alone cannot be used by female participants/female partners of male participants to prevent pregnancy).

ii. Male participants must ensure effective contraception for at least 12 weeks after the last dose of STZ that includes at least one barrier method.

Exclusion Criteria:

1. Circumstances that raise doubt about free, unconstrained consent to study participation (e.g. in a prisoner or mentally handicapped person)
2. Poor general condition where delay in treatment cannot be tolerated or death within three months is likely.
3. Poor social condition which would make it unlikely that the patient would be able to complete follow-up
4. The patient is pregnant or breast-feeding.
5. The patient is infected with HIV with a cluster of differentiation (CD) 4 count <220 cells/mm3. If >220 cells/mm3, patients will be included only if any of the following is applicable:

   * The patient is antiretroviral (ARV) naïve and able to postpone commencing HIV treatment for 2 months after the trial has started and then restrict regimens to those containing dolutegravir (see section 12.6.2 on ARVs) or The patient is ARV experienced (has been on ARV´s a minimum of 5 months) and able to switch to a dolutegravir-based regimen.
   * Nucleosidic reverse transcriptase inhibitors are permitted as concomitant medication.
   * Protease inhibitors as part of antiretroviral treatment regimens: need to be stopped at least 3 days before the start of study treatment (WK00, d1) for a patient to be eligible.
   * Efavirenz as part of antiretroviral treatment regimens: may not be taken during 14 days before the start of study treatment (WK00, d1) for a patient to be eligible.
6. The patient has a known intolerance to any of the study drugs or concomitant disorders or conditions for which study drugs or standard TB treatment are contraindicated.
7. The patient has a history of, or current evidence of clinically relevant cardiovascular metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy, or any other condition that will influence treatment response, study adherence or survival in the judgement of the investigator, especially:

   1. Conditions or history that predispose to epileptic seizures: personal or first-degree family history of epileptic seizures, stroke or transient ischemic attack, or history of severe traumatic head or brain injury, or meningitis/encephalitis, or others
   2. Neuropathy, or significant psychiatric disorder like depression or schizophrenia; especially if treatment for those has ever been required or is anticipated to be required
   3. Clinically significant evidence of severe TB (e.g. miliary TB, TB meningitis, but not limited lymph node involvement)
   4. Serious lung conditions other than TB, or significant respiratory impairment in the discretion of the investigator
   5. Any diabetes mellitus
   6. Cardiovascular disease such as myocardial infarction, heart failure, coronary heart disease, arrhythmia, tachyarrhythmia, or pulmonary hypertension
   7. Arterial hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure of ≥90 mmHg on two occasions during screening).
   8. Long QT syndrome or family history of long QT syndrome or sudden death of unknown or cardiac-related cause
   9. Alcohol or other drug abuse that is sufficient to significantly compromise the safety or cooperation of the patient, that includes substances prohibited by the protocol or has led to significant organ damage at the discretion of the investigator.
8. Any of the following laboratory findings at screening:

   1. Serum amino aspartate transferase (AST) and/or alanine aminotransferase (ALT) activity >3x the upper limit of normal (ULN),
   2. serum alkaline phosphatase or y-glutamyl transferase > 2.5x the ULN,
   3. serum total bilirubin level >1.5x the ULN
   4. estimated creatinine clearance (eCrCl; using the Cockcroft and Gault formula (52) lower than 30 ml/min
   5. serum albumin < 2.8 mg/dl
   6. haemoglobin level <7.0 g/dl
   7. platelet count <50,000/mm3,
   8. serum potassium below the lower level of normal for the laboratory
   9. serum creatine phosphokinase > 5x ULN
   10. blood glucose at screening of less than 70mg/dL (3.9mmol/L)
9. ECG findings in the screening ECG: (one or more):

   1. Fridericia corrected QT (QTcF) interval of >0.450 s
   2. Atrioventricular (AV) block with PR interval > 0.20 s,
   3. QRS complex > 120 milliseconds
   4. any other changes in the ECG that are clinically relevant as per discretion of the investigator
10. Restricted medication:

    1. Treatment with any other investigational drug within 1 month prior to enrolment or enrolment into other clinical (intervention) trials during participation.
    2. Previous anti-TB treatment with drugs active against Mycobacterium tuberculosis (MTB) within the last 3 months.
    3. Unable or unwilling to abide by the requirements regarding restricted medication or have taken restricted medication. Restricted medication includes the following drug classes:

       * anti-TB drugs
       * medication that lowers the threshold for epileptic seizures
       * medication that prolongs the QTcF interval
       * drugs that affect monoamineoxidase or serotonin metabolism
       * CYP 450 inhibitors or inducers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Change in sputum mycobacterial load over time | Days 01 - 84
  Change in mycobacterial load over time on treatment as quantified by change in time to positivity in BD MGIT 960® liquid culture.
Primary safety endpoint: proportion of patients experiencing adverse events as defined below | Days 01 - 98
  * Proportion of adverse events of Grade 3 severity or higher
  * Proportion of adverse events possibly, probably or definitely related to study drugs
  * Proportion of treatment discontinuations or interruptions related to adverse events/serious adverse events
  * Specific ECG endpoints:
    * Frequency, severity and type of ECG alterations
    * Changes to PR, RR, QRS, QT, Fridericia-corrected QT [QTcF]
    * Proportion of participants with QTcF > 500ms on treatment
    * Proportion of participants with a prolongation of QTcF > 60ms relative to baseline measurement

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint 1: Time to stable culture conversion | Days 01 - 98
  Time to stable culture conversion to negative on liquid media (defined as two negative cultures without an intervening positive culture)
Secondary Efficacy Endpoint 2: Culture conversion in liquid media | Days 01 - 98
  Proportion of participants converting to negative sputum culture in liquid media (defined as two negative cultures without an intervening positive culture) at each time point during treatment
Secondary Efficacy Endpoint 3: Culture conversion on solid media | Days 01 - 98
  Proportion of participants converting to negative sputum culture on solid media at WK 08
Secondary Efficacy Endpoint 4: No conversion to negative culture | Days 01 - 98
  Proportion of participants not converting to negative culture, and participants developing drug resistance
Pharmacokinetics Endpoint Sutezolid 1: AUC 0-24 | Day 14
  A PK analysis of STZ and its main metabolite will be carried out from 7 different blood samples on day 14 by measuring the STZ-plasma concentration and creating an area under the plasma concentration curve from morning dosing to 24 hours after
Pharmacokinetics Endpoint Sutezolid 2: Cmax | Day 14
  A PK analysis of STZ and its main metabolite will be carried out from 7 different blood samples on day 14 by measuring the STZ-plasma concentration and defining the observed maximum concentration of STZ on day 14
Pharmacokinetics Endpoint Sutezolid 3: Tmax | Day 14
  A PK analysis of STZ and its main metabolite will be carried out from 7 different blood samples on day 14 by measuring the STZ-plasma concentration and defining the time to reach maximum concentration of STZ on day 14
Pharmacokinetics Endpoint Sutezolid 4: Cmin | Day 14
  A PK analysis of STZ and its main metabolite will be carried out from 7 different blood samples on day 14 by measuring the STZ-plasma concentration and defining the observed minimum concentration of STZ on day 14
Pharmacokinetics Endpoint Sutezolid 5: Cl/F | Day 14
  A PK analysis of STZ and its main metabolite will be carried out from 7 different blood samples on day 14 by measuring the STZ-plasma concentration and defining the apparent oral clearance of STZ on day 14
Pharmacokinetics Endpoint Sutezolid 6: Vd/F | Day 14
  A PK analysis of STZ and its main metabolite will be carried out from 7 different blood samples on day 14 by measuring the STZ-plasma concentration and defining the apparent volume of distribution of STZ on day 14
Pharmacokinetics Endpoint Sutezolid 7: t1/2 | Day 14
  A PK analysis of STZ and its main metabolite will be carried out from 7 different blood samples on day 14 by measuring the STZ-plasma concentration and defining the terminal half-life time of STZ on day 14
Pharmacokinetics Endpoint Midazolam | Days -1 and 14
  PK probe drug/CYP 3A4 enzyme induction endpoint: ratio of midazolam area under the curve (AUC) 0-24 (RAUC) at days -1, and day 14 (in arm 5 only)
Pharmacokinetics Endpoint Bedaquiline | Days 7, 14, 28, 56 and 84
  Bedaquiline (BDQ) Cmin at 5 time points during treatment, comparing arms 1 and 5.
Exploratory endpoint 1: rate of change in MBLA | Days 01 - 98
  Exploratory endpoints will be analysed depending on laboratory capacity and budget and may not be tested in all trial sites equally.
  • Rate of change in molecular bacterial load assay (MBLA) during treatment
Exploratory endpoint 2: time to negative MBLA | Days 01 - 98
  Exploratory endpoints will be analysed depending on laboratory capacity and budget and may not be tested in all trial sites equally.
  • Time to stable conversion to negative MBLA (defined as two negative MBLAs without an intervening positive).
Exploratory endpoint 3: time to stable culture conversion in MBLA | Days 01 - 98
  Exploratory endpoints will be analysed depending on laboratory capacity and budget and may not be tested in all trial sites equally.
  • Time to stable culture conversion to negative in MBLA (defined as two negative MBLAs without an intervening positive)
Exploratory endpoint 4: rate of change in bacterial load | Days 01 - 98
  Exploratory endpoints will be analysed depending on laboratory capacity and budget and may not be tested in all trial sites equally.
  • Rate of change in bacterial load measured by quantification of sputum lipoarabinomannan (LAM) during treatment
Mycobacterial Identification and Characterization Endpoint 1: MIC | Days 01 - 98
  Sputum cultures grown from the screening period, and the last sputum sample with mycobacterial growth will be assessed as follows:
  • Minimum inhibitory concentrations (MIC) of BDQ, Delamanid (DLM), Moxifloxacin (MXF), STZ.
Mycobacterial Identification and Characterization Endpoint 2: mutations | Days 01 - 98
  Sputum cultures grown from the screening period, and the last sputum sample with mycobacterial growth will be assessed as follows:
  • Frequency of acquired mutations in the infecting strain over treatment assessed by whole genome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, Prof., Study Director — University Hospital, LMU Munich, Division of Infectious Diseases and Tropical Medicine
Locations (4):
- The Aurum Institute for Health Research, Johannesburg, South Africa
- Tanzania (3):
  - Kilimanjaro Clinical Research Institute, Moshi, Arusha
  - Ifakara Health Institute, Bagamoyo
  - National Institute for Medical Research (NIMR - MMRC), Mbeya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinrich N, Manyama C, Koele SE, Mpagama S, Mhimbira F, Sebe M, Wallis RS, Ntinginya N, Liyoyo A, Huglin B, Minja LT, Wagnerberger L, Stoycheva K, Zumba T, Norena I, Peter DD, Makkan H, Sloan DJ, Brake LT, Schildkraut J, Aarnoutse RE, McHugh TD, Wildner L, Boeree M, Aldana BH, Phillips PPJ, Hoelscher M, Svensson EM; PanACEA consortium. Sutezolid in combination with bedaquiline, delamanid, and moxifloxacin for pulmonary tuberculosis (PanACEA-SUDOCU-01): a prospective, open-label, randomised, phase 2b dose-finding trial. Lancet Infect Dis. 2025 Nov;25(11):1208-1218. doi: 10.1016/S1473-3099(25)00213-0. Epub 2025 Jul 8. PMID 40645196